CLINICAL TRIAL: NCT07308418
Title: The Influence of Vibrotactile Stimulation on Self-selected Walking Speed in People With Parkinson's Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Magnes AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-01560
Record Dates: First submitted 2025-12-01; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-11

CONDITIONS: Parkinson's Disease (PD)
Keywords: Parkinson's Disease; Gait analysis; Vibrotactile feedback
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vibrotactile feedback while walking (Active Comparator)
  Interventions: Device: Vibrotactile feedback during walking

INTERVENTIONS:
Device: Vibrotactile feedback during walking — NUSHU smart shoes give real time gait feedback during walking.

SUMMARY:
The study tests whether a smart shoe (NUSHU) that provides vibrotactile stimulation can improve walking speed in people with Parkinson's disease. Sixteen participants complete two short walking tests-with and without vibration-to compare gait speed, cadence, stride length, usability, and safety. It is a low-risk pilot study meant to generate first evidence for future research.

DETAILED DESCRIPTION:
Study Overview

This monozentric, prospective within-subject crossover pilot study investigates whether vibrotactile stimulation provided by the NUSHU, a CE-certified smart shoe, can influence spatiotemporal gait parameters-primarily self-selected walking speed-in adults with Parkinson's disease (PD). Parkinson's disease is often associated with reduced gait speed, shorter strides, and altered cadence, all of which are clinically relevant because they correlate with morbidity, fall risk, and quality of life.

Rationale

Earlier research suggests that vibration can positively influence gait by modulating proprioception, but existing devices have been impractical or clinically cumbersome. The NUSHU integrates sensors and vibration modules into an everyday shoe, enabling precise, phase-specific stimulation during the swing phase. Since no previous PD studies have tested this device, the project seeks to assess feasibility, safety, and initial efficacy signals.

Participants

Sixteen adults with a confirmed Parkinson's diagnosis will be recruited from multiple Physiozentrum Zürich locations. Key inclusion requirements include stable medication, ability to walk ≥ 200 m without resting, and sufficient understanding of German. Exclusion criteria include neuropathy, atypical parkinsonism, major comorbid gait disorders, or cognitive impairment that may interfere with procedures.

Study Design and Procedures

Participants attend a single 45-minute session consisting of:

Informed consent and eligibility assessment

Instruction on NUSHU use

Two 2-minute walking tests (with and without vibration), in randomized order

A 15-minute washout between tests

Completion of the System-Usability-Scale (SUS) questionnaire

Continuous monitoring and documentation of safety events and perceived stability

The assessor is blinded regarding the stimulation condition to reduce bias.

Outcomes

Primary outcome:

Difference in self-selected gait speed between vibration vs. no-vibration conditions.

Secondary outcomes:

* Cadence
* Stride length
* Usability (SUS-DE)
* Safety observations and subjective stability ratings

Statistics As an exploratory pilot, the study is not powered for confirmatory conclusions. Paired statistical tests (t-test or Wilcoxon) will evaluate within-subject differences. Descriptive methods and Bonferroni-corrected secondary analyses will complement the primary evaluation.

Ethics & Risk Classified as Risk Category A, the study involves minimal risk, mainly the normal risk associated with walking. Strict inclusion criteria and supervised testing aim to reduce fall risk. Data will be pseudonymized and securely stored. Although participants receive no direct clinical benefit, the findings will support future research on technology-assisted mobility strategies for PD.

Purpose:

* Overall, the study aims to understand:
* The short-term effect of vibrotactile stimulation on gait
* The feasibility, usability, and safety of NUSHU in a PD population
* Whether larger, controlled trials are justified

ELIGIBILITY:
Inclusion criteria:

* A medically confirmed diagnosis of Parkinson's disease on the physiotherapy prescription.
* Stable medication for at least four weeks (no change in dopaminergic therapy).
* The ability to walk at least 200 metres without stopping.
* Minimum age: 18 years
* Sufficient knowledge of German to understand the study information and complete the questionnaires.
* Written informed consent form

Exclusion criteria:

* Atypical or secondary Parkinsonism
* Sensory disturbances in the feet (e.g. polyneuropathy).
* Other neurological, orthopaedic or internal medical conditions that significantly affect walking
* Cognitive impairments that interfere with understanding the study information or following instructions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change in self-selected walking speed (m/s) | Once during 120 seconds
  Change in self-selected walking speed (m/s), measured over a 2-minute walking test with and without stimulation by the NUSHU. Walking speed is measured in m/s as a continuous metric variable, which is an objective and established way of measuring walking speed. The calculation is performed by dividing the total distance covered by the time in seconds (120 seconds).
Change in self-selected gait speed | One visit of 45 minutes

IPD SHARING:
Plan to Share IPD: No